CLINICAL TRIAL: NCT04443660
Title: Autophagy/Apoptosis Balance During Pregnancy
Acronym: GROSSAUTOP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2019-01/SB-01
Record Dates: First submitted 2020-06-04; First posted 2020-06-23 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Pregnancy Related
Keywords: Autophagy; Apoptosis
MeSH Terms: interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum and mononuclear blood cells
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group A: without medical history or risk factors, with a normal pregnancy
  Interventions: Other: Blood test
- Group B: without medical history or risk factors, developing a pregnancy complication
  Interventions: Other: Blood test
- Group C: with risk of complication, having a normal pregnancy
  Interventions: Other: Blood test
- Group D: with a risk of complication, developing a pregnancy complication
  Interventions: Other: Blood test

INTERVENTIONS:
Other: Blood test — Blood samples taken to test levels of autophagy and apoptosis

SUMMARY:
The object of this study is to assess the intra- and inter-individual variability of apoptosis and autophagy activities in women during pregnancy: 1 / in women with a normal pregnancy and 2 / in pregnant women particularly at risk of complications.

The study investigators hypothesize that there would be an intra-trophoblastic dialogue between the mechanisms of autophagy and apoptosis, the promotion of one partially inhibiting the other. The increase in trophoblastic autophagy during pregnancy could thus constitute an anti-apoptosis defense phenomenon, the exhaustion of which would lead to cellular apoptosis and to pathogenic consequences when it devastates the syncytiotrophoblast.

ELIGIBILITY:
Inclusion Criteria:

* Patients followed at the CHU Nimes prior to 33 weeks gestation who give birth at the hospital
* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan

Exclusion Criteria:

* The subject is participating in a category 1 interventional study associated with a medication, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Multiple pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All pregnant women followed at the Nimes University Hospital for their pregnancy. Patients will be recruited among those consulting hospital gynecologists from the 3rd month of pregnancy but also through the circuit of specific gynecology-obstetrics consultations receiving in particular women with a history and / or risk factors for pathological pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-04-07 (Actual)

PRIMARY OUTCOMES:
Potential autophagy induction activity in all groups | Day 0
  Microtubule-associated protein 1A/1B-light chain 3 fluorescence ratio
Potential autophagy induction activity in all groups | Month 1
  Microtubule-associated protein 1A/1B-light chain 3 fluorescence ratio
Potential autophagy induction activity in all groups | Month 2
  Microtubule-associated protein 1A/1B-light chain 3 fluorescence ratio
Potential autophagy induction activity in all groups | Month 3
  Microtubule-associated protein 1A/1B-light chain 3 fluorescence ratio
Potential autophagy induction activity in all groups | Month 4
  Microtubule-associated protein 1A/1B-light chain 3 fluorescence ratio
Potential autophagy induction activity in all groups | Month 5
  Microtubule-associated protein 1A/1B-light chain 3 fluorescence ratio
Potential autophagy induction activity in all groups | Delivery plus or minus 2 weeks (Month 6)
  Microtubule-associated protein 1A/1B-light chain 3 fluorescence ratio

SECONDARY OUTCOMES:
Type of autophagy inhibition per patient in all groups | Day 0
  Early/late; measured by microtubule-associated protein 1A/1B-light chain 3 fluorescence ratio
Type of autophagy inhibition per patient in all groups | Month 1
  Early/late; measured by microtubule-associated protein 1A/1B-light chain 3 fluorescence ratio
Type of autophagy inhibition per patient in all groups | Month 2
  Early/late; measured by microtubule-associated protein 1A/1B-light chain 3 fluorescence ratio
Type of autophagy inhibition per patient in all groups | Month 3
  Early/late; measured by microtubule-associated protein 1A/1B-light chain 3 fluorescence ratio
Type of autophagy inhibition per patient in all groups | Month 4
  Early/late; measured by microtubule-associated protein 1A/1B-light chain 3 fluorescence ratio
Type of autophagy inhibition per patient in all groups | Month 5
  Early/late; measured by microtubule-associated protein 1A/1B-light chain 3 fluorescence ratio
Type of autophagy inhibition per patient in all groups | Delivery plus or minus 2 weeks (Month 6)
  Early/late; measured by microtubule-associated protein 1A/1B-light chain 3 fluorescence ratio
Potential apoptosis induction activity in all groups | Day 0
  % cells positive for Annexin V
Potential apoptosis induction activity in all groups | Month 1
  % cells positive for Annexin V
Potential apoptosis induction activity in all groups | Month 2
  % cells positive for Annexin V
Potential apoptosis induction activity in all groups | Month 3
  % cells positive for Annexin V
Potential apoptosis induction activity in all groups | Month 4
  % cells positive for Annexin V
Potential apoptosis induction activity in all groups | Month 5
  % cells positive for Annexin V
Potential apoptosis induction activity in all groups | Delivery plus or minus 2 weeks (Month 6)
  % cells positive for Annexin V
Inter- and intra-individual apoptosis/autophagy ratio in all groups | Day 0
Inter- and intra-individual apoptosis/autophagy ratio in all groups | Month 1
Inter- and intra-individual apoptosis/autophagy ratio in all groups | Month 2
Inter- and intra-individual apoptosis/autophagy ratio in all groups | Month 3
Inter- and intra-individual apoptosis/autophagy ratio in all groups | Month 4
Inter- and intra-individual apoptosis/autophagy ratio in all groups | Month 5
Inter- and intra-individual apoptosis/autophagy ratio in all groups | Delivery plus or minus 2 weeks (Month 6)
Autophagy kinetics between groups | Day 0
  measured by microtubule-associated protein 1A/1B-light chain 3 fluorescence ratio
Autophagy kinetics between groups | Month 1
  measured by microtubule-associated protein 1A/1B-light chain 3 fluorescence ratio
Autophagy kinetics between groups | Month 2
  measured by microtubule-associated protein 1A/1B-light chain 3 fluorescence ratio
Autophagy kinetics between groups | Month 3
  measured by microtubule-associated protein 1A/1B-light chain 3 fluorescence ratio
Autophagy kinetics between groups | Month 4
  measured by microtubule-associated protein 1A/1B-light chain 3 fluorescence ratio
Autophagy kinetics between groups | Month 5
  measured by microtubule-associated protein 1A/1B-light chain 3 fluorescence ratio
Autophagy kinetics between groups | Delivery plus or minus 2 weeks (Month 6)
  measured by microtubule-associated protein 1A/1B-light chain 3 fluorescence ratio
Apoptosis kinetics between groups | Day 0
  measured by % cells positive for Annexin V
Apoptosis kinetics between groups | Month 1
  measured by % cells positive for Annexin V
Apoptosis kinetics between groups | Month 2
  measured by % cells positive for Annexin V
Apoptosis kinetics between groups | Month 3
  measured by % cells positive for Annexin V
Apoptosis kinetics between groups | Month 4
  measured by % cells positive for Annexin V
Apoptosis kinetics between groups | Month 5
  measured by % cells positive for Annexin V
Apoptosis kinetics between groups | Delivery plus or minus 2 weeks (Month 6)
  measured by % cells positive for Annexin V
Placental Growth Factor in each group | Day 0
  pg/ml measured by ELISA
Placental Growth Factor in each group | Month 1
  pg/ml measured by ELISA
Placental Growth Factor in each group | Month 2
  pg/ml measured by ELISA
Placental Growth Factor in each group | Month 3
  pg/ml measured by ELISA
Placental Growth Factor in each group | Month 4
  pg/ml measured by ELISA
Placental Growth Factor in each group | Month 5
  pg/ml measured by ELISA
Placental Growth Factor in each group | Delivery plus or minus 2 weeks (Month 6)
  pg/ml measured by ELISA
Soluble fms-like tyrosine kinase-1 | Day 0
  pg/ml measured by ELISA
Soluble fms-like tyrosine kinase-1 | Month 1
  pg/ml measured by ELISA
Soluble fms-like tyrosine kinase-1 | Month 2
  pg/ml measured by ELISA
Soluble fms-like tyrosine kinase-1 | Month 3
  pg/ml measured by ELISA
Soluble fms-like tyrosine kinase-1 | Month 4
  pg/ml measured by ELISA
Soluble fms-like tyrosine kinase-1 | Month 5
  pg/ml measured by ELISA
Soluble fms-like tyrosine kinase-1 | Delivery plus or minus 2 weeks (Month 6)
  pg/ml measured by ELISA
Constitutive thrombophilia | Day 0
  presence/absence of the prothrombin gene or factor V Leiden mutation, protein S, C or antithrombin deficiency
Acquired thrombophilia | Day 0
  Presence/absence of anti-phospholipid antibodies (lupus anticoagulant and/or anti beta2-GP1 and/or anti-cardiolipid).
Acquired thrombophilia | Month 1
  Presence/absence of anti-phospholipid antibodies (lupus anticoagulant and/or anti beta2-GP1 and/or anti-cardiolipid).
Acquired thrombophilia | Month 2
  Presence/absence of anti-phospholipid antibodies (lupus anticoagulant and/or anti beta2-GP1 and/or anti-cardiolipid).
Acquired thrombophilia | Month 3
  Presence/absence of anti-phospholipid antibodies (lupus anticoagulant and/or anti beta2-GP1 and/or anti-cardiolipid).
Acquired thrombophilia | Month 4
  Presence/absence of anti-phospholipid antibodies (lupus anticoagulant and/or anti beta2-GP1 and/or anti-cardiolipid).
Acquired thrombophilia | Month 5
  Presence/absence of anti-phospholipid antibodies (lupus anticoagulant and/or anti beta2-GP1 and/or anti-cardiolipid).
Acquired thrombophilia | Delivery plus or minus 2 weeks (Month 6)
  Presence/absence of anti-phospholipid antibodies (lupus anticoagulant and/or anti beta2-GP1 and/or anti-cardiolipid).
Whole blood count | Day 0
Whole blood count | Month 1
Whole blood count | Month 2
Whole blood count | Month 3
Whole blood count | Month 4
Whole blood count | Month 5
Whole blood count | Delivery plus or minus 2 weeks (Month 6)
Renal function | Day 0
  creatinemia, proteinuria / creatinuria ratio
Renal function | Month 1
  creatinemia, proteinuria / creatinuria ratio
Renal function | Month 2
  creatinemia, proteinuria / creatinuria ratio
Renal function | Month 3
  creatinemia, proteinuria / creatinuria ratio
Renal function | Month 4
  creatinemia, proteinuria / creatinuria ratio
Renal function | Month 5
  creatinemia, proteinuria / creatinuria ratio
Renal function | Delivery plus or minus 2 weeks (Month 6)
  creatinemia, proteinuria / creatinuria ratio
Fibrin levels | Day 0
  D dimers and fibrin monomers
Fibrin levels | Month 1
  D dimers and fibrin monomers
Fibrin levels | Month 2
  D dimers and fibrin monomers
Fibrin levels | Month 3
  D dimers and fibrin monomers
Fibrin levels | Month 4
  D dimers and fibrin monomers
Fibrin levels | Month 5
  D dimers and fibrin monomers
Fibrin levels | Delivery plus or minus 2 weeks (Month 6)
  D dimers and fibrin monomers
Inflammation | Day 0
  C-reactive protein level
Inflammation | Month 1
  C-reactive protein level
Inflammation | Month 2
  C-reactive protein level
Inflammation | Month 3
  C-reactive protein level
Inflammation | Month 4
  C-reactive protein level
Inflammation | Month 5
  C-reactive protein level
Inflammation | Delivery plus or minus 2 weeks (Month 6)
  C-reactive protein level
Activated partial thromboplastin time | Day 0
  seconds
Activated partial thromboplastin time | Month 1
  seconds
Activated partial thromboplastin time | Month 2
  seconds
Activated partial thromboplastin time | Month 3
  seconds
Activated partial thromboplastin time | Month 4
  seconds
Activated partial thromboplastin time | Month 5
  seconds
Activated partial thromboplastin time | Delivery plus or minus 2 weeks (Month 6)
  seconds
Prothrombin time | Day 0
  seconds
Prothrombin time | Month 1
  seconds
Prothrombin time | Month 2
  seconds
Prothrombin time | Month 3
  seconds
Prothrombin time | Month 4
  seconds
Prothrombin time | Month 5
  seconds
Prothrombin time | Delivery plus or minus 2 weeks (Month 6)
  seconds
Fibrinogen level | Day 0
  g/L
Fibrinogen level | Month 1
  g/L
Fibrinogen level | Month 2
  g/L
Fibrinogen level | Month 3
  g/L
Fibrinogen level | Month 4
  g/L
Fibrinogen level | Month 5
  g/L
Fibrinogen level | Delivery plus or minus 2 weeks (Month 6)
  g/L
Thrombin generation time | Month 1
  seconds
Thrombin generation time | Month 2
  seconds
Thrombin generation time | Month 3
  seconds
Thrombin generation time | Month 4
  seconds
Thrombin generation time | Month 5
  seconds
Thrombin generation time | Delivery plus or minus 2 weeks (Month 6)
  seconds
Thrombin generation time | Day 0
  seconds
fetal haemoglobin | Month 1
  g/L
fetal haemoglobin | Month 2
  g/L
fetal haemoglobin | Month 3
  g/L
fetal haemoglobin | Month 4
  g/L
fetal haemoglobin | Month 5
  g/L
fetal haemoglobin | Delivery plus or minus 2 weeks (Month 6)
  g/L

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Bouvier, Principal Investigator — CHU Nimes
Locations (1):
- CHU de Nimes, Nîmes, France

REFERENCES:
- [Result] Fortier M, Portes M, Demattei C, Nouvellon E, Mercier E, Bourguignon C, Chea M, Gris JC, Letouzey V, Bouvier S. Thrombin generation reference values using the ST Genesia and STG-Thromboscreen assay in pregnant women. Thromb Res. 2026 Jan;257:109558. doi: 10.1016/j.thromres.2025.109558. Epub 2025 Nov 29. No abstract available. PMID 41371090